CLINICAL TRIAL: NCT00474916
Title: A Phase 2 Double-Blind Dose Escalation Study of KRN5500 for Neuropathic Pain in Patients With Cancer
Brief Title: Neuropathic Pain in Patients With Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DARA Therapeutics (Industry)
Responsible Party: Linda Jett, MSN, Clinical Director, DARA BioSciences and DARA Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DTCL100
Record Dates: First submitted 2007-05-15; First posted 2007-05-17 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic pain; Cancer
MeSH Terms: conditions — Neuralgia; Neoplasms | interventions — KRN 5500

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KRN5500 (Experimental): KRN5500 escalating dose of .6, 1.2, 1.8, or 2.2 mg/m2 in IV infusion of normal saline
  Interventions: Drug: KRN5500
- Normal Saline (Placebo Comparator): Placebo consists of IV infusion of normal saline
  Interventions: Drug: KRN5500; Drug: Placebo

INTERVENTIONS:
Drug: KRN5500 — Patients are seen weekly and dosed for pain with IV medication of active drug/KRN5500 or placebo . The dose can be escalated, from .6 mg/m2, to 1.2, 1.8, and 2.2 mg/m2.
Drug: Placebo — Normal Saline given as dose escalation for placebo
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to collect beginning information on whether intravenous (IV) administration of KRN5500 is safe and effective for treatment of neuropathic pain in patients with cancer.

DETAILED DESCRIPTION:
Neuropathic pain is a type of pain that results from nerve damage and is characterized by an abnormal hypersensitivity to harmless as well as harmful stimuli. This type of pain is extremely difficult to manage, fails to respond to standard analgesic medications or interventions, and often gets worse instead of better over time. Current approved therapeutic agents often have intolerable side effects and limited efficacy. Thus, there is an urgent need to develop safe and effective drugs to treat neuropathic pain.

Study DTCL100 will be conducted at multiple centers and will enroll patients that have advanced cancer AND neuropathic pain that has not responded well to previous treatment. Eighteen patients will be randomly assigned to receive up to 8 doses of active drug (KRN5500) or placebo. A maximum of 8 doses will be administered weekly over a 10 week period. Patients are encouraged to complete at least 4 treatment visits before a decision is made to complete the full 10 weeks of treatment and the 1 month followup period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of advanced or recurrent cancer
* No options for curative chemotherapy, but palliative chemotherapy allowed under certain conditions
* Refractory neuropathic pain rated 4 or greater on 0-10 scale and failure to respond to 2 commonly used treatments
* If taking opioids for pain, stable regimen over past week before enrolling
* Karnofsky performance status of 40 or more
* Females must be sterile or post-menopausal

Exclusion Criteria:

* Radiation to site of neuropathic pain for past 4 weeks
* Major surgery within past 2 weeks
* Liver function and other key labs outside normal parameters
* ECG showing significant abnormality
* Myocardial Infarction (heart attack) within past 6 months
* History of interstitial lung disease
* History of severe allergic reaction to drugs containing polysorbate 80
* Other investigational drug within 2 weeks or 5 half-lives (whichever is longer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-06; Primary Completion 2009-03 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Average pain intensity over the previous 24 hours as measured by a numeric rating scale (NRS) ranging from 0 to 10 where 0 represents "no pain" and 10 represents the "worst possible pain." | Weekly for 10 weeks plus 30 day followup

SECONDARY OUTCOMES:
Physical Examination, Vital signs and body weight, Electrocardiogram, Laboratory parameters, Adverse events, Clinical Opiate Withdrawal Scale, rescue medication, Proportion of patients who achieved a 33% reduction in pain intensity | Weekly for 10 weeks plus 30 day followup

CONTACTS AND LOCATIONS:
Overall Officials: Richard Penson, MD, MRCP, Principal Investigator — Massachusetts General Hospital
Locations (12):
- United States (11):
  - Cancer Institute Medical Group, Los Angeles, California
  - Ghassan Al-Jazayrly, M.D., Inc., Los Angeles, California
  - University of California / Irvine Chao Family Comprehensive Cancer Center, Orange, California
  - Keog Pharma, Inc., Jupiter, Florida
  - Hematology and Oncology Specialists, LLC, Covington, Louisiana
  - St. Agnes Healthcare, Inc, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - East Orange VA Medical Center, East Orange, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Carolina Pain Institute, PA, Winston-Salem, North Carolina
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Dr. Rivera-Colon, Rio Piedras, Puerto Rico